CLINICAL TRIAL: NCT03408028
Title: Therapeutic Intervention Code in a Cognitive Geriatric Unit: Retrospective Analysis
Brief Title: Therapeutic Intervention Code in a Cognitive Geriatric Unit
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of Clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB- status code
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Cognitive Impairment
Keywords: Therapeutic code; Geriatry
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive impairment: Geriatric patients with a cognitive impairment
  Interventions: Other: Medical File consultation

INTERVENTIONS:
Other: Medical File consultation — Medical File consultation

SUMMARY:
The diagnostic and therapeutic progresses, associated with modifications in lifestyle and socio-cultural level of populations, have led to a remarkable increase in life expectancy. At the same time, the increasing medicalization of the individual has eroded the traditional boundaries between health and illness, normal and pathological state. This leads to the patient losing his sense of ownership of his own death. If most patients died at home before the Second World War, 75% of the population dies in hospital or institution at the present date.

Most hospitals and care institutions have developed codes, in multidisciplinary internal consultation, to address the interruption or lack of implementation of treatments that make no sense from a medical point of vue. This avoids therapeutic relentlessness.The code in place within the CHU Brugmann is:

* code A: no therapeutic restriction
* code B: not to be resuscitated
* code C: not to be intensively treated (no escalation in therapeutic treatments)
* code D: best palliative care (progressive de-escalation in therapeutic treatments).

These codes are established in consultation with the patient or his legal representative and are re-evaluated in a multidisciplinary way every week.

Planning a care path and therefore establishing a therapeutic code is particularly important for people with cognitive impairment and dementia because the progressive loss of cognitive abilities complicates the process of decision making.

A large part of the admissions are made via the emergency department. For these patients, no therapeutic plan has been established beforehand. However, the perception of the functional and cognitive status of the patient directly influences the intensity of care provided. Cognitive disorders are a risk factor for the exclusion of access to palliative care for the elderly patient.

The objectives of this study are:

* To establish a record of the therapeutic limitation codes in an acute cognitive geriatric unit
* To correlate the therapeutic limitation code with the comorbidities of the patients

ELIGIBILITY:
Inclusion Criteria:

Elderly patients with cognitive impairment admitted in the geriatric unit 83 within the CHU Brugmann between 01-01-2016 and 31-12-2016.

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Eldelry patients with cognitive imparement admitted in the geriatric unit 83 within the CHU Brugmann between 01-01-2016 and 31-12-2016.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Therapeutic code | From 01-01-2016 till 31-12-2016
  Therapeutic code
Cumulative Illness Rating Scale for Geriatrics | From 01-01-2016 till 31-12-2016
  This scoring system measures the chronic medical illness ("morbidity") burden while taking into consideration the severity of chronic diseases in 14 items representing individual body systems. The cumulative final score can theoretically vary from 0 to 56.

SECONDARY OUTCOMES:
Age | From 01-01-2016 till 31-12-2016
  Age
Sex | From 01-01-2016 till 31-12-2016
  Sex
Ethnicity | From 01-01-2016 till 31-12-2016
  Ethnicity

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Natalia Grande Pérez, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No